CLINICAL TRIAL: NCT01338324
Title: Protocol for Correlating Enteropathic Severity and Small Intestinal CYP3A4 Activity in Patients With Celiac Disease
Acronym: Cyp
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Govind K Makharia, Dr. Govind K Makharia, All India Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: N-1229
Record Dates: First submitted 2011-04-06; First posted 2011-04-19 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Celiac Disease
Keywords: Biomarker; Pharmacokinetics; Villous; Simvastatin; Celiac disease
MeSH Terms: conditions — Celiac Disease | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 20 mg single dose on day 1

SUMMARY:
The small bowel biopsy is the cornerstone of for the diagnosis of celiac disease. In addition to being the gold standard for the initial diagnosis of celiac disease, periodic biopsies are also recommended on an ongoing basis for this life-long disease. However, biopsy evaluation is invasive and expensive. Therefore, there is a need for simple, non-invasive tests that can be performed on celiac patients with subclinical disease.

The present study is based on the hypothesis that the expression and activity of cytochrome P450 CYP3A4 in the small intestinal mucosa is a sensitive measure of enteropathy. Therefore small intestinal CYP3A4 activity will be markedly different in celiac disease patients with active disease as compared to patients in remission. Small intestinal CYP3A4 activity will be measured in three ways:

(i) Cmax of oral simvastatin, a widely used drug that is predominantly metabolized by small intestinal CYP3A4; (ii) AUC of oral simvastatin; and (iii) Measurement of CYP3A4 activity in two small bowel biopsies.

DETAILED DESCRIPTION:
The proposed study is based on the hypothesis that the expression and activity of cytochrome P450 CYP3A4 in the small intestinal mucosa is a sensitive measure of enteropathy. Therefore small intestinal CYP3A4 activity will be markedly different in celiac disease patients with active disease as compared to patients in remission. Small intestinal CYP3A4 activity will be measured in three ways:

(iv) Cmax of oral simvastatin, a widely used medication that is predominantly metabolized by small intestinal CYP3A4; (v) AUC of oral simvastatin; and (vi) Measurement of CYP3A4 activity in two small bowel biopsies.

Objectives Primary Objectives

* To test the hypothesis that a positive correlation exists between villus height: crypt depth (Vh:Cd) ratio and the specific activity of CYP3A4 in small intestinal biopsy samples derived from subjects with celiac disease.
* To test the hypothesis that an inverse correlation exists between small intestinal villus height: crypt depth (Vh:Cd) ratio and the maximum serum concentration (Cmax) of simvastatin (20 mg, orally dosed after fasting) in subjects with celiac disease

Secondary Objectives:

* To test the hypothesis that an inverse correlation exists between small intestinal villus height: crypt depth (Vh:Cd) ratio and the serum area-under-the-curve (AUC) of simvastatin (20 mg, orally dosed after fasting) in subjects with celiac disease
* To test the hypothesis that a positive correlation exists between small intestinal villus height : crypt depth (Vh:Cd) ratio and the relative expression level of CYP3A4 protein in subjects with celiac disease.
* To test the hypothesis that an inverse correlation exists between small intestinal villus height : crypt depth (Vh:Cd) ratio and the concentration of simvastatin (20 mg, orally dosed after fasting) in a 6-hour urine collection from subjects with celiac disease.
* To test the hypothesis that a positive correlation exists between villus height : crypt depth (Vh:Cd) ratio and the specific activity of CYP3A4 in small intestinal biopsy samples derived from subjects with celiac disease who have followed a gluten-free diet for > 1 year.
* To test the hypothesis that an inverse correlation exists between small intestinal villus height: crypt depth (Vh:Cd) ratio and the maximum serum concentration (Cmax) of simvastatin (20 mg, orally dosed after fasting) in subjects with celiac disease who have followed a gluten-free diet for > 1 year.
* To test the hypothesis that an inverse correlation exists between small intestinal villus height: crypt depth (Vh:Cd) ratio and the serum area-under-the-curve (AUC) of simvastatin (20 mg, orally dosed after fasting) in subjects with celiac disease who have followed a gluten-free diet for > 1 year.
* To test the hypothesis that a positive correlation exists between serum anti-transglutaminase antibody levels and the specific activity of CYP3A4 in small intestinal biopsy samples derived from subjects with celiac disease.
* To test the hypothesis that a positive correlation exists between the average daily consumption of dietary gluten and the specific activity of CYP3A4 in small intestinal biopsy samples derived from subjects with celiac disease.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort A: Suspected celiac sprue patients who have:

   (i) Positive Anti-transglutaminase IgA levels.

   (ii) Either a first-degree relative with diagnosed celiac sprue or at least one of the following symptoms:

   iron deficiency, osteopenia, chronic diarrhea.
2. Cohort B: Diagnosis of celiac disease confirmed by medical history,

   (i)Histology of small intestinal mucosa on small bowel biopsy and elevated serum concentrations of anti-transglutaminase antibodies.

   (ii)Followed gluten-free diet for at least 1 year.
3. If the subject is female, she is eligible to enter and participate in this study if she is physiologically incapable of becoming pregnant or has a negative urine pregnancy test at screening.

Exclusion Criteria:

1. Smoking
2. Any gastrointestinal or hepatic disease besides celiac sprue.
3. Clinically significant renal disease.
4. Use of any prescription or non-prescription drugs (including vitamins and herbal supplements) must be discontinued 30 days prior to study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax ) of simvastatin (20 mg, orally dosed after fasting) in subjects with celiac sprue | 12 hours

SECONDARY OUTCOMES:
Duodenal level of cytochrome CYP3A4 | 72 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr Govind K Makharia, MD, DM, DNB, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India